CLINICAL TRIAL: NCT01581853
Title: Pilot Simplification Study to Lopinavir/Ritonavir 800/200 mg Monotherapy Regimen Once Daily
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Podzamczer (Other)
Responsible Party: Sponsor-Investigator, Daniel Podzamczer, MD. HIV/AIDS Program Director. HIV Unit. Infectious Disease Service, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMON; 2011-005981-39 (EudraCT Number)
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2013-04

CONDITIONS: HIV
Keywords: HIV; AIDS; MONOTHERAPY; PILOT; LOPINAVIR/RITONAVIR
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lopinavir/ritonavir 800 mg / 200mg (Other): Kaletra 200/50 mg comprimidos recubiertos con película Lopinavir/ritonavir 800 mg / 200mg will be changed from its approved posology (2 times daily)to once daily in patients with undetectable viral load and in stable treatment with Lopinavir/ritonavir 800 mg / 200mg in monotherapy for at least 6 months
  Interventions: Drug: Lopinavir/ritonavir 800 mg / 200mg

INTERVENTIONS:
Drug: Lopinavir/ritonavir 800 mg / 200mg — Lopinavir/ritonavir 800 mg / 200mg will be change from its approved posology (2 times daily)to once daily in patients with undetectable viral load and in stable treatment with Lopinavir/ritonavir 800 mg / 200mg in monotherapy for at least 6 months
  Other Names: Kaletra 200/50 mg comprimidos recubiertos con película

SUMMARY:
Lopinavir/ritonavir monotherapy is currently a well known and widely used strategy, while Lopinavir/ritonavir 800/200 mg once a day in a triple-therapy was approved a few years ago. The purpose of this study is to evaluate efficacy and safety of Lopinavir/ritonavir 800/200 mg monotherapy once a day.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18, HIV positive
* Patients receiving a monotherapy regimen (Lopinavir/ritonavir twice daily)during the last 6 months
* Undetectable viral load (<40 copies/ml) during the last 6 months
* Patients that accept participation in the study and sign the Informed Consent Form
* Childbearing females with negative pregnancy tests and using appropriate contraceptive measures

Exclusion Criteria:

* Opportunistic disease, cancer or any other active disease with specific treatment
* Active addiction to illegal drugs or active use of psychotropic drugs
* Mental retardation diagnosis, or mental dementia or severe psychiatric disorder (excluding major depression disorder solved > 3 months)
* Females who are breastfeeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
plasma viral load <40 copies/mL | Week 48
  HIV Plasma Viral Load <40 copies/ml at week 48.

SECONDARY OUTCOMES:
Stability in the plasma levels of Lopinavir/ritonavir during all study visits | Weeks 4, 8, 12, 16, 24, 36 and 48
  Determination of plasma concentrations of the study drug at weeks 4, 8, 12, 16, 24, 36 and 48
Tolerability | Weeks 4, 8, 12, 16, 24, 36 and 48
  Possible Adverse Events will be collected in all study visits and laboratory tests will also be performed in all study visits (weeks 4, 8, 12, 16, 24, 36 and 48)
Adherence | Weeks 4, 8, 12, 16, 24, 36 and 48
  Medication adherence will be evaluated in all the study visits after making a reconciliation of the medication dispensed and returned by the patients
Satisfaction | Weeks 4, 8, 12, 16, 24, 36 and 48
  Patients' satisfaction with the new regimen will be evaluated using a questionnaire (SMAQ)
- Efficacy in CSF | At least 4 weeks on study treatment
  - In a subsample of patients (10) HIV-1 RNA in CSF will be assessed (added as per amendment)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Podzamczer, MD, Principal Investigator — Hospital Universitari de Bellvitge; Hernando Knobel, MD, Principal Investigator — Hospital del Mar
Locations (2):
- Spain (2):
  - Hospital del Mar, Bercelona, Barcelona
  - Hospital Universitary de Bellvitge, L'Hospitalet de Llobregat, Barcelona